CLINICAL TRIAL: NCT01176578
Title: Exercise Training, CACs, and Vascular Function in Older Veterans With IGT (Impaired Glucose Tolerance)
Brief Title: Exercise Endothelial Progenitor Cells (EPCs) and Type 2 Diabetes
Acronym: EPC-DM
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Baltimore VA Medical Center (U.S. Federal Agency)
Collaborators: University of Maryland, Baltimore (Other)
Responsible Party: Principal Investigator, Steven J. Prior, Ph.D., Assistant Professor, Baltimore VA Medical Center
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: HP-00047188
Record Dates: First submitted 2010-08-05; First posted 2010-08-06 (Estimated); Last update posted 2025-09-19 (Actual); Status verified 2025-09

CONDITIONS: Type 2 Diabetes Mellitus
MeSH Terms: conditions — Diabetes Mellitus, Type 2

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- T2DM (Experimental): Type 2 Diabetes Mellitus
  Interventions: Other: Aerobic Exercise Training
- IGT (Experimental): Impaired Glucose Tolerance
  Interventions: Other: Aerobic Exercise Training
- NGT (Active Comparator): Normal Glucose Tolerance
  Interventions: Other: Aerobic Exercise Training

INTERVENTIONS:
Other: Aerobic Exercise Training — 6 months of aerobic exercise training, 3 days per week

SUMMARY:
The discovery of the role of endothelial progenitor cells (EPCs) and their involvement in the cardiovascular complications of type 2 diabetes (T2DM) would quickly have a significant impact on the millions of Americans who have T2DM. This project is designed to 1) determine the mechanisms underlying EPC dysfunction in older, sedentary adults with T2DM compared those with normal glucose metabolism and impaired glucose metabolism, and 2) determine if aerobic exercise training is an efficacious therapy for EPC dysfunction in T2DM, and whether improvement in EPC number and function translates to improved endothelial function, increased capillarization, and improved glucose metabolism in T2DM.

ELIGIBILITY:
Inclusion Criteria:

* Age 50-80
* Non-smoker
* If woman, postmenopausal >1 year

Exclusion Criteria:

* History of heart disease or stroke
* Cancer
* Poorly controlled hypertension or dyslipidemia
* Kidney or Liver diseases

Ages: 50 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 70 (Estimated)
Dates: Start 2011-07 (Actual); Primary Completion 2021-12-31 (Actual); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Endothelial progenitor cell number | Baseline
Endothelial progenitor cell number | 6-month
Skeletal muscle capillarization | Baseline
Skeletal muscle capillarization | 6-month

SECONDARY OUTCOMES:
Cardiorespiratory Fitness | Baseline
Cardiorespiratory Fitness | 6-month

CONTACTS AND LOCATIONS:
Locations (1):
- Baltimore VA Medical Center, Baltimore, Maryland, United States